CLINICAL TRIAL: NCT00642395
Title: Velcade®-Melphalan Association as Conditioning Regimen Before Autologous Stem-cell Transplantation in Multiple Myeloma Patients Under 65 Years
Brief Title: Velcade®-Melphalan Association in Autologous Stem-Cell Transplantation (ASCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Intergroupe Francophone du Myelome (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0603603
Record Dates: First submitted 2008-03-13; First posted 2008-03-25 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Autologous Stem Cells Transplantation; High Dose Melphalan; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): bortézomib
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — bortezomib-Melphalan
  Other Names: Velcade

SUMMARY:
Intensification with autologous stem cell (ASCT) is currently the most effective treatment for subjects under 65 and the essential goal is to achieve complete response (CR) or very good partial response (VGPR= greater than 90% reduction of monoclonal component). However, only 50% of patients achieve this CR/VGPR even with tandem ASCT early in the course of disease.

Optimization of the conditioning regimen could improve this CR/VGPR rate. The combinaison of Velcade and HD Melphalan has never been evaluated. However, at conventional doses, Velcade potentiates the antimyeloma effect of Melphalan without inducing any common toxicity.

This study will be conducted in patients under the age of 65 with de novo multiple myeloma or in first relapse, with Salmon and Durie stage of III, II, I with one symptomatic bone lesion (radiological)and no contraindication to intensification. The primary objective will be to increase the CR/VGPR rate 3 months after autologous peripheral blood stem cell transplantation conditioned by Velcade-Melphalan from 40% to 70%. With alpha=5% and bêta=10%, 61 patients will be included.

Secondary objectives will be to assess the toxicity of the Velcade-Melphalan conditioning regimen, the progression-free survival and the overall survival after intensification. Response rates will be evaluated according to the response criteria defined by. Analysis will be performed on an intention-to-treat basis.

After conventional induction therapy and PBSC collection, patients will be offered this new conditioning regimen. they will be free to refuse this regimen, in which case they will receive standard intensification therapy by Melphalan 200 mg/m² followed by autologous stem cell transplantation.

Evaluation will occur at 3 months post intensification.

ELIGIBILITY:
Inclusion Criteria:

At time of diagnosis

* De novo multiple myeloma patients under 65 or in first relapse, in whom screening for chromosome 13 deletion and beta2microglobulin assay have been performed.
* Salmon and Durie Stage: III, II, I with symptomatic bone lesion (radiological)
* Patient's written informed consent
* No clinical signs of heart failure or coronary insufficiency with LVEF>50%
* No hepatic in insufficiency: bilirubin<35μmol/l and SGOT, SGPT, alkaline phosphatase less than 2.5 N
* No respiratory insufficiency: normal pulmonary function tests and DLCO>50%
* No pre-existing renal impairment not related to the disease
* No history of any other malignant disease with the exception of basal cell carcinoma and stage I cervical cancer
* Negative HIV serology
* Effective contraception when justified

At the time of transplantation

* Good performance status (WHO score≤2)
* Creatinine≤170μmol/l and no ineligibility criteria for intensification
* Stem cells harvest ≥ 5x10E6 CD34/kg for 2 ASCT
* Absence of progressive disease before transplantation

Exclusion Criteria:

* Known refusal of the subject to participate to the study
* Female subject who is pregnant or breast-feeding
* History of allergy to any of the study medications, their analogues, or excipients in the various formulations
* Main liver insufficiency
* ≥ Grade 3 peripheral neuropathy on clinical examination within 14 days before enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the Complete Response and Very Good Partial Response (VGPR) rates 3 months after autologous blood stem cell transplantation conditioned by Velcade-Melphalan | 3 months after autologous stem cell transplantation

SECONDARY OUTCOMES:
Assess the toxicity of this Velcade-Melphalan conditioning regimen (hematological and visceral toxicity-NCI criteria) - To assess the progression-free survival after transplantation - To assess the overall survival after tran | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Murielle ROUSSEL, MD, Principal Investigator — Purpan Hospital - UH Toulouse
Locations (34):
- France (34):
  - Service of Blood Deseases - South Hospital, Amiens
  - Service of Clinical Hematology - Bocage Hospital, Angers
  - Service of Clinical Hematology - Cote Basque Hospital, Bayonne
  - Service of Clinical Hematology - Minjoz Hospital, Besançon
  - Service of Clinical Hematology - Avicenne Hospital, Bobigny
  - Service of Clinical Hematology - A. Morvan Hospital, Brest
  - Service of Clinical Hematology - F. Baclesse Center, Caen
  - Service of Clinical Hematology - Army Instruction Hospital of Percy, Clamart
  - Service of Clinical Hematology - UH of Clermont-Ferrand, Clermont-Ferrand
  - Service of Oncohematology - Louis Pasteur Hospital, Colmar
  - Service of Hematology - Bocage Hospital, Dijon
  - Service of Hematology - General Hospital, Dunkirk
  - Service of Hematology - A. Michallon Hospital, Grenoble
  - Service of Hematology - Claude Hurriez Hospital, Lille
  - Service of Hematology - Léon Bérard Center, Lyon
  - Service of Hematology - Edouard Herriot Hospital, Lyon
  - Service of Hematology - Lyon Sud Hospital, Lyon
  - Service of Hematology - Paoli Calmette Institute, Marseille
  - Service of Hematology - Notre Dame du Bon Secours Hospital, Metz
  - Service of Blood Deseases - UH of Nantes, Nantes
  - Service of Clinical Hematology - Archet 1 Hospital, Nice
  - Service of Oncology - Archet 1 Hospital, Nice
  - Service of Hematology - Hotel Dieu, Paris
  - Service of Hematology - Cochin Hospital, Paris
  - Service of Blood Deseases - Saint Antoine Hospital, Paris
  - Service of Hematology - Jean Bernard Hospital, Poitiers
  - Service of Hematology - R.Debré Hospital, Reims
  - Service of Hematology - Pontchaillou Hospital, Rennes
  - Service of Hematology -Henri Becquerel Center, Rouen
  - Service of Hematology - Hautepierre Hospital, Strasbourg
  - Service of Clinical Hematology - Purpan hospital TSA 40031, Toulouse
  - Service of Onco-Hematology - Bretonneau Hospital, Tours
  - Service of Hematology - Brabois Hospital, Vandœuvre-lès-Nancy
  - Service of Hematology -Gustave Roussy Institute, Villejuif

REFERENCES:
- [Result] Roussel M, Moreau P, Huynh A, Mary JY, Danho C, Caillot D, Hulin C, Fruchart C, Marit G, Pegourie B, Lenain P, Araujo C, Kolb B, Randriamalala E, Royer B, Stoppa AM, Dib M, Dorvaux V, Garderet L, Mathiot C, Avet-Loiseau H, Harousseau JL, Attal M; Intergroupe Francophone du Myelome (IFM). Bortezomib and high-dose melphalan as conditioning regimen before autologous stem cell transplantation in patients with de novo multiple myeloma: a phase 2 study of the Intergroupe Francophone du Myelome (IFM). Blood. 2010 Jan 7;115(1):32-7. doi: 10.1182/blood-2009-06-229658. Epub 2009 Nov 2. PMID 19884643